CLINICAL TRIAL: NCT04292158
Title: The New Golden Standard: the Early Warning Score Algorithm
Acronym: EAGLE
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Collaborators: Academisch Ziekenhuis Maastricht (Other); KU Leuven (Other); Ziekenhuis Oost-Limburg (Other); Hasselt University (Other); Maastricht University (Other)
Responsible Party: Principal Investigator, Patrizio Lancellotti, Professor, University of Liege
Other Study IDs: 2018/184
Record Dates: First submitted 2019-10-01; First posted 2020-03-02 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Early Warning Score
Keywords: Early warning score; Vital parameters; Predictive algorithm; Medical Devices

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Main Group: Hospitalized for at least 1 day clinic stay at the participating hospitals
  Interventions: Device: SomnoTouch; Device: MOX

INTERVENTIONS:
Device: SomnoTouch — The patient will be equipped with the SomnoTouch device. This device is able to record and estimate the following data:
  ECG data PPG data Heart rate Respiration rate Blood pressure (mmHg) Oxygen saturation (%).
  All patient will be stored for further analysis.
Device: MOX — The patient will be equipped with the MOX device. This device is able to record and estimate the following data:
  Accelerometers data Activity Body posture
  All patient will be stored for further analysis.

SUMMARY:
The objective is this study is the development and implementation of a smart algorithm to compute an early warning indicator able to predict early patient deterioration.

DETAILED DESCRIPTION:
Data will be collected at the three sites using the SomnoTouchTM and MOXTM devices, commercially available and CE approved. Every month, the data will be sent to the KUL and UM to develop the algorithm. Study centers will also send some pre-defined patient characteristics extracted from the patient's EMR to better contextualize the data.

The EWS formula has a free interpretation of the vital parameters weighting and the vital parameters to be taken into account in the scoring system. Therefore, many variants of the EWS arose the past decade (i.e. MEWS, NEWS). The algorithm developed in this study should define an objective approach for the EWS formula, diminishing the discordances regarding the weight per parameter. Using a patient-personalized approach, the definite algorithm should be based on the patient's vital parameter measured during his/her whole hospitalization, generating a patient-personalized weight per parameter and an overall reliable EWS scoring system.

The EWS score is often only measured twice per day per patient, creating a large window for disease worsening. The algorithm developed in this study could be deployed along the wearable device developed in the WearIT4Health project. The device would continuously feed the algorithm with data acquired from its sensors. Thus, the EWS would be computed every 10 seconds.

The EWS scoring system has already been proven to be an effective approach in reducing clinical deterioration, reducing the admission to intensive care units and thus overall reducing mortality. However, as mentioned above the EWS is measured in a rather low frequency. Therefore, estimation of the EWS score via continuous monitored parameters should further increase patient survival.

The primary objective of the EAGLE study is to collect continuously monitored vital and activity parameter data and use it to develop an algorithm that can early identify clinical deterioration to optimize the application of the EWS system.

ELIGIBILITY:
Exclusion Criteria:

* Suffering from infectious disease
* Participating to another study that could intervene with the study results (e.g. experimental medication that could affect the heart rate).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospitalized for at least 1 day at the participating hospitals excluding patients admitted at high intensity units: Intensive care units, Coronary care units, Emergency room.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Precision of predictive early warning score algorithm | Up to 1 week
  Precision defined of truepositives divided by the sum of truepositives and truenegatives. This measure indicates how often the predictive EWS was right in identifying adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Patrizio Lancellotti, Principal Investigator — Liège University Hospital - CHU de Liège; Pierre Delanaye, Study Director — Liège University Hospital - CHU de Liège; Arnaud Ancion, Study Director — Liège University Hospital - CHU de Liège; Pieter Vandervoort, Study Director — Department of Cardiology and Department Future Health, Ziekenhuis Oost-Limburg; Dianne de Korte-de Boer, Study Chair — Maastricht University Medical Centre, department of Anesthesiology
Locations (3):
- Belgium (2):
  - Ziekenhuis Oost-Limburg, Genk, Limbourg
  - Centre Hospitalier Universitaire de Liège, Liège
- Maastricht University Medical Center+, Maastricht, Netherlands

REFERENCES:
- [Background] Gerry S, Birks J, Bonnici T, Watkinson PJ, Kirtley S, Collins GS. Early warning scores for detecting deterioration in adult hospital patients: a systematic review protocol. BMJ Open. 2017 Dec 3;7(12):e019268. doi: 10.1136/bmjopen-2017-019268. PMID 29203508
- [Background] Jarvis S, Kovacs C, Briggs J, Meredith P, Schmidt PE, Featherstone PI, Prytherch DR, Smith GB. Aggregate National Early Warning Score (NEWS) values are more important than high scores for a single vital signs parameter for discriminating the risk of adverse outcomes. Resuscitation. 2015 Feb;87:75-80. doi: 10.1016/j.resuscitation.2014.11.014. Epub 2014 Nov 26. PMID 25433295
- [Background] Moon A, Cosgrove JF, Lea D, Fairs A, Cressey DM. An eight year audit before and after the introduction of modified early warning score (MEWS) charts, of patients admitted to a tertiary referral intensive care unit after CPR. Resuscitation. 2011 Feb;82(2):150-4. doi: 10.1016/j.resuscitation.2010.09.480. Epub 2010 Nov 5. PMID 21056524
- [Background] Ajami S, Teimouri F. Features and application of wearable biosensors in medical care. J Res Med Sci. 2015 Dec;20(12):1208-15. doi: 10.4103/1735-1995.172991. PMID 26958058
- [Background] Smith MEB, Chiovaro JC, O'Neil M, Kansagara D, Quinones A, Freeman M, Motu'apuaka M, Slatore CG. Early Warning System Scores: A Systematic Review [Internet]. Washington (DC): Department of Veterans Affairs (US); 2014 Jan. Available from http://www.ncbi.nlm.nih.gov/books/NBK259026/ PMID 25506953